CLINICAL TRIAL: NCT01536496
Title: A Prospective, Randomized Comparison Of Rapid Thrombelastography (r-TEG) And Conventional Coagulation Testing For Guiding The Diagnosis And Haemostatic Resuscitation Of Trauma Patients At Risk For Post-Injury Coagulopathy
Brief Title: Comparison of Rapid Thrombelastography and Conventional Coagulation Testing for Haemostatic Resuscitation in Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Haemonetics Corporation (Industry)
Responsible Party: Principal Investigator, Ernest E. Moore, MD, Director, Surgery/Trauma Service, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COMIRB # 10-0477
Record Dates: First submitted 2011-07-19; First posted 2012-02-22 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Acute Coagulopathy
Keywords: trauma; hemorrhagic shock; thrombelastography; coagulopathy; transfusion; resuscitation
MeSH Terms: conditions — Wounds and Injuries; Shock, Hemorrhagic; Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (INR, PTT, fibrinogen, D-dimer) (Active Comparator): Patients randomized to the Control Group will receive blood component therapy guided by conventional coagulation tests per usual clinical practice. The control arm involves the use of conventional coagulation tests (aPTT, INR, fibrinogen level, D-dimer) to diagnose and describe post-injury coagulopathy and to guide blood product replacement. In the Control Group, blood will be drawn for conventional coagulation testing (aPTT, INR, platelet count, fibrinogen level, D-dimer) at Baseline (as defined above), then twice more during the first six hours at the discretion of the treating team, then again at 12 hours and at 24 hours post-injury. The current institutional massive transfusion protocol will be followed. Only the results pertinent to the group to which randomized will be released to the treating team, unless otherwise requested.
  Interventions: Biological: Blood product transfusion based on conventional coagulation tests.
- Test (r-TEG) (Active Comparator): Patients randomized to the r-TEG guided haemostatic resuscitation group (Test Group) will receive blood component therapy per usual clinical practice. The test arm involves the use of rapid-TEG to diagnose and describe post-injury coagulopathy and to guide blood product replacement per institutional algorithm. In the Test Group, blood for r-TEG will be collected on admission, or upon entering the operating room, depending on the acuity of the injury (Baseline), and this will be followed by two additional r-TEG analyses during the first six hours at the discretion of the treating team (attending surgeon, anesthesiologist) and then two further r-TEG analyses at 12 hours and at 24 hours post-injury respectively. The current institutional massive transfusion protocol will be followed. Only the results pertinent to the group to which randomized will be released to the treating team, unless otherwise requested.
  Interventions: Biological: Blood product transfusion based on rapid thrombelastography (r-TEG) results.

INTERVENTIONS:
Biological: Blood product transfusion based on conventional coagulation tests. — Transfusion of blood products.
  Arms: Control (INR, PTT, fibrinogen, D-dimer)
Biological: Blood product transfusion based on rapid thrombelastography (r-TEG) results. — Transfusion of blood products.
  Arms: Test (r-TEG)

SUMMARY:
The purpose of this study is to compare rapid thrombelastography (r-TEG) with conventional coagulation testing for diagnosing and treating coagulation abnormalities in severely injured patients who are likely to require transfusion therapy.

DETAILED DESCRIPTION:
This is a prospective, randomized study comparing rapid thrombelastography (r-TEG) with conventional coagulation testing for diagnosing post-injury coagulopathy and guiding haemostatic resuscitation strategy in severely injured patients arriving at the trauma center who are likely to require transfusion therapy.

Our global hypothesis is that:

1. r-TEG is an effective tool for early identification of specific coagulation abnormalities via real time analysis, providing rapid results at the point of care (POC),
2. r-TEG can be used to guide resuscitation strategy by permitting transfusion based upon individual patient deficits,
3. r-TEG will result in appropriate transfusion of plasma, cryoprecipitate, and platelets in the individual trauma patient,
4. r-TEG will result in reduced transfusion requirements in patients with post-injury coagulopathy.

Our specific study aims are:

1. To compare r-TEG parameters [TEG-ACT, alpha angle, K value, MA (maximum amplitude), G value (clot strength), and fibrinolysis (EPL=estimated percent lysis)] with conventional coagulation testing [aPTT, INR, platelet count, fibrinogen level, D-dimer] in their ability to diagnose and monitor coagulation abnormalities in the trauma patient specifically.
2. To compare blood product administration (packed red blood cells, fresh frozen plasma, cryoprecipitate and apheresis platelets) in the first 24 hours post-injury when transfusion is guided by r-TEG versus conventional coagulation tests.
3. To determine whether normalization of r-TEG values predicts cessation of coagulopathic bleeding better than normalization of conventional clinical coagulation tests based upon clinical impressions of the treating surgeons and review of operative records and outcome.
4. To determine and compare patterns of transfusion ratios of packed red blood cells: fresh frozen plasma: platelets for resuscitation of patients with post-injury coagulopathy in the r-TEG versus conventional coagulation test guided groups for the first 24 hours post-injury.
5. To determine and compare the timeframes of blood product administration throughout the first 24 hours post-injury when transfusion is guided by r-TEG versus conventional coagulation testing.
6. To compare the incidence of hemorrhage-related deaths as: very early mortality (<2 hours post-injury), early (2<6 hours post-injury) and delayed (6-24 post-injury) based upon review of death/autopsy records for date, time and cause of death in patients whose resuscitation is guided by r-TEG versus conventional coagulation testing.
7. To compare a) the incidence of transfusion associated lung injury (TRALI), transfusion associated circulatory overload (TACO), acute respiratory distress syndrome (ARDS), and multiple organ failure (MOF); b) the length of stay in the surgical intensive care unit (SICU) and the number of ventilator free days in the SICU; and c) late mortality (>24 hour to Day 30), including day number and cause of death, in patients whose resuscitation is guided by r-TEG versus conventional coagulation testing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age >18 years admitted to Denver Health Medical Center.
2. Blunt or penetrating trauma sustained < 6 hours before admission, with Injury Severity Score > 15 (ISS>15), likely to require transfusion of RBC within 6 hours from admission as indicated by clinical assessment.

Exclusion Criteria:

1. Age < 18 years.
2. Documented chronic liver disease (total bilirubin >2.0 mg/dL). Advanced cirrhosis discovered on laparotomy will be a criterion for study withdrawal and exclusion of conventional coagulation or r-TEG/TEG data from the analysis).
3. Known inherited defects of coagulation function (e.g. hemophilia, Von Willebrand's disease).
4. Prisoner.
5. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest E. Moore, M.D., Principal Investigator — Denver Health
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 09/25/2010 and the last one was enrolled on 03/21/2014. The patients were enrolled when they met the inclusion criteria for the study, which were the criteria that activate the massive transfusion protocol. Enrollment occured upon arrival either in Emergency Room or in Operating Room.
Groups:
- Test (r-TEG): Patients randomized to the r-TEG guided haemostatic resuscitation group (Test Group) will receive blood component therapy per usual clinical practice. The test arm involves the use of rapid-TEG to diagnose and describe post-injury coagulopathy and to guide blood product replacement per institutional algorithm. In the Test Group, blood for r-TEG will be collected on admission, or upon entering the operating room, depending on the acuity of the injury (Baseline), and this will be followed by two additional r-TEG analyses during the first six hours at the discretion of the treating team (attending surgeon, anesthesiologist) and then two further r-TEG analyses at 12 hours and at 24 hours post-injury respectively. The current institutional massive transfusion protocol will be followed. Only the results pertinent to the group to which randomized will be released to the treating team, unless otherwise requested.
  Blood product transfusion based on rapid thrombelastography (r-TEG) results.:
Period: Overall Study
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Started | 57 | 57
Completed | 55 | 56
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG) | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [25 to 55] | 41 [28 to 54] | 39 [28 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 33
  Male | 41 | 37 | 78
Injury Severity Score (ISS) [Median (Inter-Quartile Range); unit: Scores on a scale] — 0 to 75, higher score means worse outcome
  Scores on a scale | 33 [25 to 43] | 29.5 [23 to 41] | 30 [24 to 43]
Base Deficit (BD) [Median (Inter-Quartile Range); unit: mEq/L] — Base deficit refers to lack of bases in the blood. Bases are crucial in sustaining the acid-base homeostasis in the human body. Base deficit is an indicator of metabolic component of blood pH, as opposed to carbon dioxide, which is an indicator of respiratory component of blood pH. Base deficit outside of normal values (-2 to 2 mEq/L) usually means a shift in homeostasis towards acids or metabolic acidosis. More negative values are indicative of more profound disturbance in homeostasis.
  mEq/L | 13.7 [9 to 18] | 11.0 [9 to 16] | 12.0 [9 to 18]
International Normalized Ratio (INR) [Median (Inter-Quartile Range); unit: units on a scale] — The reference range of the local clinical laboratory is 0.83-1.19. A high INR indicates a higher risk of bleeding, while a low INR suggests a higher risk of developing a clot.
  units on a scale | 1.46 [1.2 to 2.3] | 1.45 [1.2 to 1.7] | 1.45 [1.2 to 1.9]
Platelet count [Median (Inter-Quartile Range); unit: k/uL] — The reference range of the local clinical laboratory is 150-400 k/uL.
  k/uL | 214 [165 to 279] | 214 [145 to 318] | 214 [150 to 291]
Fibrinogen [Median (Inter-Quartile Range); unit: mg/dL] — The reference range of the local clinical laboratory is 200.0-485.0 mg/dL.
  mg/dL | 113 [68 to 139] | 132 [94 to 240] | 122 [75 to 201]
D-dimer [Median (Inter-Quartile Range); unit: ug/mL] — The reference range of the local clinical laboratory is <0.50 ug/mL.
  ug/mL | 12.9 [6 to 20] | 10.3 [2 to 20] | 11.1 [4 to 20]
TEG ACT (activated clotting time) [Median (Inter-Quartile Range); unit: seconds] — The reference range of the local clinical laboratory is 78.0-110.0.
  seconds | 128 [113 to 278] | 128 [113 to 140] | 128 [113 to 195]
TEG Angle [Median (Inter-Quartile Range); unit: degrees] — The reference range of the local clinical laboratory is 66.0-82.0 degrees.
  degrees | 50.9 [28 to 69] | 52.3 [30 to 70] | 51.5 [29 to 69]
TEG MA (maximal amplitude) [Median (Inter-Quartile Range); unit: mm] — The reference range of the local clinical laboratory is 54.0-72.0 mm.
  mm | 47.5 [34 to 53] | 53.9 [28 to 63] | 50.9 [31 to 60]
TEG LY30 [Median (Inter-Quartile Range); unit: percent of clot lysis at 30 minutes] — The reference range of the local clinical laboratory is 0.0-7.4%. Percent of clot lysis 30 minutes after maximal amplitude (MA) was finalized.
  percent of clot lysis at 30 minutes | 0.5 [0 to 4.4] | 1.2 [0.1 to 4.2] | 0.9 [0 to 4.3]

OUTCOME MEASURES:

1. Primary Outcome: 28 Day In-hospital Mortality
Time Frame: 28 days in hospital
Measure: Number; unit: participants
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
participants | 20 | 11
Statistical Analysis 1: Comparison: Control (INR, PTT, Fibrinogen, D-dimer) vs Test (r-TEG); Chi-square test; Test type: Superiority or Other; p = 0.04, Chi-squared

2. Secondary Outcome: Deaths Specified as Early Mortality (<6 Hours Post-injury) and Delayed Mortality (6-24 Hours Post-injury).
Time Frame: Within 24 hours post-injury.
Measure: Number; unit: deaths
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
deaths
  Number of deaths <6 hours from injury | 12 | 4
  Number of deaths 6-24 hours from injury | 8 | 7

3. Secondary Outcome: Deaths Related to Coagulopathic Bleeding Based Upon Clinical Impressions of the Treating Surgeons and Review of Operative Records and Outcome (Hours Since Injury).
Time Frame: Up to 28 days post-injury.
Measure: Number; unit: deaths
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
deaths | 11 | 5

4. Secondary Outcome: Time to Death From Injury in Hours.
Time Frame: From time of injury to 28th day of hospitalization.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 20 | 11
hours | 4.2 [1.2 to 9.9] | 10.4 [4.5 to 200.3]

5. Secondary Outcome: Change in INR Test Results.
Description: A high International Normalized Ratio (INR) indicates a higher risk of bleeding, while a low INR suggests a higher risk of developing a clot.
Time Frame: Within first 6 hours post-injury, 12 and 24 hours post-injury.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Control (INR, PTT, Fibrinogen, D-dimer): Patients randomized to the Control Group will receive blood component therapy guided by conventional coagulation tests per usual clinical practice. The control arm involves the use of conventional coagulation tests (INR, fibrinogen level, D-dimer) to diagnose and describe post-injury coagulopathy and to guide blood product replacement. In the Control Group, blood will be drawn for conventional coagulation testing (INR, platelet count, fibrinogen level, D-dimer) at Baseline (as defined above), then twice more during the first six hours at the discretion of the treating team, then again at 12 hours and at 24 hours post-injury. The current institutional massive transfusion protocol will be followed. Only the results pertinent to the group to which randomized will be released to the treating team, unless otherwise requested.
  Blood product transfusion based on conventional coagulation tests.: Transfusion of blood products.
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
units on a scale
  INR at 6 hours | 1.5 [1.3 to 2.2] | 1.8 [1.3 to 2.1]
  INR at 12 hours | 1.4 [1.2 to 1.6] | 1.4 [1.3 to 1.9]
  INR at 24 hours | 1.5 [1.4 to 1.7] | 1.4 [1.3 to 2]

6. Secondary Outcome: Change in Fibrinogen Test Results.
Time Frame: Within first 6 hours post-injury, 12 and 24 hours post-injury.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Control (INR, Fibrinogen, D-dimer): Patients randomized to the Control Group will receive blood component therapy guided by conventional coagulation tests per usual clinical practice. The control arm involves the use of conventional coagulation tests (INR, fibrinogen level, D-dimer) to diagnose and describe post-injury coagulopathy and to guide blood product replacement. In the Control Group, blood will be drawn for conventional coagulation testing (INR, platelet count, fibrinogen level, D-dimer) at Baseline (as defined above), then twice more during the first six hours at the discretion of the treating team, then again at 12 hours and at 24 hours post-injury. The current institutional massive transfusion protocol will be followed. Only the results pertinent to the group to which randomized will be released to the treating team, unless otherwise requested.
  Blood product transfusion based on conventional coagulation tests.: Transfusion of blood products.
Arm/Group | Control (INR, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
mg/dL
  fibrinogen at 6 hours | 161.5 [112 to 175] | 153 [111 to 180]
  fibrinogen at 12 hours | 185.5 [159 to 232] | 159 [111 to 214]
  fibrinogen at 24 hours | 233 [218 to 256] | 203 [150 to 266]

7. Secondary Outcome: Change in Platelet Count Test Results.
Time Frame: Within first 6 hours post-injury, 12 and 24 hours post-injury.
Measure: Median (Inter-Quartile Range); unit: k/uL
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
k/uL
  platelet count at 6 hours | 90 [60 to 144] | 100 [89 to 140]
  platelet count at 12 hours | 116 [75 to 157] | 110 [90 to 139]
  platelet count at 24 hours | 96.5 [72 to 128] | 109 [91 to 130]

8. Secondary Outcome: Change in D-dimer Test Results.
Time Frame: Within first 6 hours post-injury, 12 and 24 hours post-injury.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
ug/mL
  D-dimer at 6 hours | 8.3 [1 to 15] | 8.7 [2 to 13]
  D-dimer at 12 hours | 8 [2 to 13] | 6.4 [3 to 13]
  D-dimer at 24 hours | 5.4 [2 to 13] | 5 [3 to 13]

9. Secondary Outcome: Change in r-TEG ACT (Activated Clotting Time) Test Results.
Time Frame: Within first 6 hours post-injury, 12 and 24 hours post-injury.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
seconds
  r-TEG ACT at 6 hours | 124 [113 to 142] | 121 [117 to 144]
  r-TEG ACT at 12 hours | 128 [121 to 144] | 121 [113 to 140]
  r-TEG ACT at 24 hours | 128 [121 to 128] | 128 [121 to 136]

10. Secondary Outcome: Change in r-TEG Angle Test Results.
Time Frame: Within first 6 hours post-injury, 12 and 24 hours post-injury.
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
degrees
  r-TEG Angle at 6 hours | 70.8 [64 to 72] | 68.2 [60 to 73]
  r-TEG Angle at 12 hours | 68.5 [60 to 70] | 65.5 [57 to 73]
  r-TEG Angle at 24 hours | 69.1 [61 to 71] | 71.3 [64 to 74]

11. Secondary Outcome: Change in r-TEG Maximal Amplitude (MA) Test Results.
Time Frame: Within first 6 hours post-injury, 12 and 24 hours post-injury.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
mm
  r-TEG MA at 6 hours | 53.8 [49 to 59] | 51 [46 to 57]
  r-TEG MA at 12 hours | 55 [52 to 57] | 56.9 [49 to 58]
  r-TEG MA at 24 hours | 56.5 [46 to 62] | 56.9 [54 to 61]

12. Secondary Outcome: Change in r-TEG LY30 Test Results.
Time Frame: Within first 6 hours post-injury, 12 and 24 hours post-injury.
Measure: Median (Inter-Quartile Range); unit: percent of clot lysis at 30 min.
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
percent of clot lysis at 30 min.
  r-TEG LY30 at 6 hours | 0 [0 to 0] | 0 [0 to 1.5]
  r-TEG LY30 at 12 hours | 0.3 [0 to 0.5] | 0.1 [0.1 to 1.5]
  r-TEG LY30 at 24 hours | 0.7 [0.2 to 1.6] | 0.7 [0.7 to 1.7]

13. Secondary Outcome: Composition and Quantity of Blood Products Transfused at 24 Hours Post-injury
Description: Amount of blood product (red blood cells, plasma, cryoprecipitate and platelets) in units.
Time Frame: 24 hours post-injury
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
units
  Red blood cell units | 11.0 [6 to 16] | 9.5 [5 to 16]
  Plasma units | 6.0 [4 to 9] | 5 [3 to 9]
  Cryoprecipitate units | 1.0 [0 to 2] | 0 [0 to 2]
  Platelet units | 1 [0 to 2] | 1 [0 to 2]

14. Secondary Outcome: Length of Stay (Days) in the Surgical Intensive Care Unit (SICU) Reported as ICU-free Days and Number of Days on the Ventialator Reported as Ventilator Free Days.
Time Frame: 28 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
days
  ICU-free days. | 8.5 [0 to 19.5] | 16 [0 to 22]
  Ventilator-free days. | 13 [0 to 22] | 18 [0 to 25]

15. Secondary Outcome: Number of Participants With Multiple Organ Failure (MOF) During This Hospitalization.
Description: Multiple Organ Failure (MOF) score (Denver method) was calculated for the participants. This score rates the dysfunction of four organ systems (pulmonary, renal, hepatic, and cardiac), which are evaluated daily throughout the patient's intensive care unit stay and graded on a scale from 0 to 3, with the total score ranging from 0-12. Higher values on the score represent worse outcome. Participants with score above 3 were considered to have MOF.
Time Frame: Up to 30 days post-injury.
Measure: Number; unit: participants
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Number analyzed (Participants) | 55 | 56
participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Up to 28 days of hospitalization.
Arm/Group | Control (INR, PTT, Fibrinogen, D-dimer) | Test (r-TEG)
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 55/55 | 56/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (INR, PTT, Fibrinogen, D-dimer) (N=55) | Test (r-TEG) (N=56)
Abnormal laboratory finding (Blood and lymphatic system disorders) | 55 (55) | 56 (56) — All subjects in this trial had abnormal lab results (coagulation, hematology, etc.) and as such were reported as adverse events to local IRB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No